CLINICAL TRIAL: NCT06462651
Title: A Double-blind, Randomised, Placebo-controlled, Parallel-group Study Evaluating the Effect of Probiotic Limosilactobacillus Reuteri (L. Reuteri) on Crying and Fussing Time in Infants With Colic
Brief Title: Effect of Probiotic Limosilactobacillus Reuteri (L. Reuteri) on Crying and Fussing Time in Infants With Colic
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: BioGaia AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CSUB0214 (CSUB0222)
Record Dates: First submitted 2024-06-12; First posted 2024-06-17 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Infantile Colic
MeSH Terms: conditions — Colic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- L. reuteri (Experimental): Dietary Supplement: L. reuteri
  Interventions: Dietary Supplement: L. reuteri
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: L. reuteri — Supplementation with drops containing L. reuteri once daily for 21 consecutive days
  Arms: L. reuteri
Dietary Supplement: Placebo — Supplementation with identical drops without L. reuteri once daily for 21 consecutive days
  Arms: Placebo

SUMMARY:
This is a double-blind, randomized, placebo-controlled, parallel-group study in infants with colic with the primary objective to evaluate crying and fussing time.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 3-12 weeks at screening.
2. Gestational age 37+0 weeks - 42+0 weeks at birth.
3. Birth weight appropriate for gestational age (AGA - weight between 10th and 90th percentile) or Large for Gestational Age (LGA - weight above the 90th percentile) determined using WHO Weight-for Age percentile guides.
4. Parents/caregivers/legal guardians are >18 years.
5. Exclusively or predominantly breastfed infants (> 50 % breast fed).
6. Willing to maintain current feeding patterns (not change formula/not change ratio of formula:breast milk etc.).
7. Readiness and the opportunity for parents/caregivers/legal guardians to fill out a study diary, questionnaires.
8. Infantile colic diagnosed according to Rome IV criteria (face-to-face consult with a physician, parents/caregivers/legal guardians must report that their infant has cried or fussed for 3 or more hours per day, during 3 or more days in the preceding week). At Visit 2, this will be confirmed by Baby's Day Diary®, at least one 24-hour period should show 3 or more hours of crying/fussing time.
9. Parents/caregivers/legal guardians with ability to understand and comply with the requirements of the study, as judged by the Investigator.
10. Parents/caregivers/legal guardians willing and able to give informed consent for their and their infant's participation in the study.
11. The mother of the infant must be willing to attend Visit 2 (Day 0), Visit 3 (Day 8), and Visit 4 (Day 22).
12. Infant is considered healthy, in the opinion of the investigator following physical exam.

Exclusion Criteria:

1. Infants with severe gastroesophageal reflux (throwing up or spitting up more than a teaspoon of milk > 8 times daily, projectile, bilious or bloody emesis).
2. Infants with failure to thrive, intrauterine growth retardation, haematochezia (blood in the stools), diarrhoea (watery stools that takes the shape of a container > 12x in breastfed and >5 in partially breastfed infants daily), or fever (38.0 degrees), as reported by parents/caregivers/ legal guardians.
3. Infants with congenital heart disease, immunodeficiency, asplenia, cancer, cystic fibrosis, and those with liver disease.
4. Infants with reported exposure to probiotics in the 7 days prior to Screening Visit (V1) and throughout the study period.
5. Infants with reported exposure to oral and/or systemic antibiotics in the 7 days prior to Screening Visit (V1) and throughout the study period.
6. Infants with reported exposure to medications, therapies, or products with the aim to relieve infantile colic including proton pump inhibitors in the 7 days prior to Screening Visit (V1) and throughout the study period.

Ages: 3 Weeks to 12 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2025-06-09 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Crying and fussing time | [Time Frame: From baseline to Day 7]
  To evaluate crying and fussing time after 7 days of supplementation with L. reuteri in infants with colic.

SECONDARY OUTCOMES:
Crying and fussing time | [Time Frame: From baseline up to Day 21]
  Change in mean daily crying and fussing time measured by Baby´s Day Diary
Crying time | [Time Frame: From baseline up to Day 21]
  Change in mean daily crying time measured by Baby´s Day Diary
Number of responders | [Time Frame: From baseline up to Day 21]
  Proportion of responders defined as reduction of daily average crying time with 50 % compared to baseline
Family quality of life (family QoL) | [Time Frame: From baseline up to Day 21]
  Change in family QoL measured by the PedsQL Family Impact Module (Acute) - Total Score
Sleeping time | [Time Frame: From baseline up to Day 21]
  Change in mean sleeping time measured by Baby´s Day Diary
Maternal depression | [Time Frame: From baseline up to Day 21]
  Change in maternal depression measured by the Edinburgh Postnatal Depression Scale Total Score

CONTACTS AND LOCATIONS:
Locations (1):
- University of Salento, University Hospital Vito Fazzi Lecce, Lecce, LE, Italy

IPD SHARING:
Plan to Share IPD: Undecided